CLINICAL TRIAL: NCT02452710
Title: Harnessing the Effect of an Open-Label Placebo on Fatigue in Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study funding was completed.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christopher Recklitis, Ph.D, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-583
Record Dates: First submitted 2015-05-19; First posted 2015-05-25 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Fatigue in Cancer Survivors
Keywords: Fatigue in Cancer Survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open-Label Placebo (Experimental): - Placebo Tablets-Twice a day for 3-4 weeks
  Interventions: Other: Placebo
- NT-Control (No Intervention): - No Placebo Tablets

INTERVENTIONS:
Other: Placebo — Open-label placebo
  Arms: Open-Label Placebo

SUMMARY:
This research study is evaluating the usefulness of a placebo (a tablet with no active ingredients) on fatigue in cancer survivors.

DETAILED DESCRIPTION:
Fatigue can be a problem for some people after cancer treatment. In clinical trials, placebos (tablets with no active ingredients) have been shown to improve symptoms of some medical conditions including fatigue. This study is being done to test the usefulness of taking placebos for improving cancer-related fatigue. In this study, the investigators are testing whether symptoms of fatigue will improve when people know they are taking a tablet with no active ingredients.

This is a randomized study, which means the participant will be put into one of two groups. Because no one knows which of the study options is best, the participant will be 'randomized' into one of the two study groups. Randomization means that the participant will be put into a group by chance. It is like flipping a coin. Neither the participant nor the research doctor will choose what group he or she will be in. The participant will have an equal chance of being placed in each of the groups.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivor, with no evidence of active disease
* ≥18 years of age
* ≥6 months and <10 years post active treatment
* Reports being bothered by fatigue in the past month and has a score of <43 on FACIT-F.
* Able to read and write in English

Exclusion Criteria:

* Being evaluated or likely to be evaluated for a medical cause of fatigue (e.g., anemia, hypothyroidism) during the study. (per provider report)
* Have indications of sleep apnea as assessed by Epworth Sleepiness scale score ≥10.
* Are receiving, or are likely to receive another intervention for the treatment of fatigue during the study period. (per provider report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue on the Functional Assessment of Cancer Therapy - Fatigue (FACIT-F) scale | Change from baseline to Day 8, and from baseline to Day 22
  13-item self-report measure of fatigue

SECONDARY OUTCOMES:
Change in Mood on the Profile of Mood Scale- Short Form (POMS-SF) | Change from baseline to Day 22
  35-items self-report mood scale
Health Related Quality of Life on the Short Form-12 (SF-12) quality of life scale | Change from baseline to Day 22
  12-item HRQOL measure
Subjective Sense of Change on fatigue, readiness for exercise and quality of life | Change from baseline to Day 8, and change from Baseline to Day 22
  3-item measure that asks participants to report changes to their level of fatigue, ability to engage in physical activity, and overall quality of life since the beginning of the research program.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Recklitis, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States